CLINICAL TRIAL: NCT00915278
Title: A Phase 1 Safety, Pharmacokinetic And Pharmacodynamic Study Of The Anti-A5B1 Integrin Monoclonal Antibody PF-04605412 Administered Intravenously To Adult Patients With Advanced Or Metastatic Solid Tumors
Brief Title: A Safety Study Of A Monoclonal Antibody Against A5B1 Integrin In Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on 26 February 2013. Risk-benefit assessment is no longer positive and does not support further development
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1001001
Record Dates: First submitted 2009-06-03; First posted 2009-06-08 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Non-Hematologic Malignancies
Keywords: Neoplasms; monoclonal antibody; PF-04605412; advanced metastatic solid tumors
MeSH Terms: conditions — Neoplasms | interventions — PF-04605412

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-04605412 (Experimental)
  Interventions: Drug: PF-04605412

INTERVENTIONS:
Drug: PF-04605412 — PF-04605412 will be administered as 2 hr IV infusion every 4 or 2 weeks. Start dose is 7.5 mg. Multiple doses are foreseen. Treatment will continue until intolerable toxicity, progression of disease or patient's refusal

SUMMARY:
Dose finding study of the MoaB PF-04605412 directed against the alpha5beta1 integrin. Main objective is to define the MTD (maximum tolerated dose) or MAD (maximum administrable dose) in cancer patients pre treated or unresponsive to standard therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced measurable or evaluable solid tumors unresponsive to currently available therapies, or for which there is no curative therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 and 1
* Life expectancy more than12 weeks
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Known brain metastasis
* Chemotherapy, radiotherapy, or any investigational cancer therapy within 4 weeks of start of screening procedures
* Major surgical procedure within 4 weeks of start of screening procedures
* Active bleeding disorder, including gastrointestinal bleeding, as evidenced by hematemesis, significant hemoptysis or melena in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (2):
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Nashville, Tennessee
- United Kingdom (3):
  - Pfizer Investigational Site, Tooting, London
  - Pfizer Investigational Site, North Cheam, Surrey
  - Pfizer Investigational Site, Sutton, Surrey

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1001001&StudyName=A%20Safety%20%20Study%20Of%20A%20Monoclonal%20Antibody%20Against%20A5B1%20Integrin%20In%20Solid%20Tumors%20

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04605412 7.5 mg: PF-04605412 7.5 mg was administered intravenously as 2 hour infusion on Day 1 of each cycle. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 11.25 mg: PF-04605412 11.25 mg was administered intravenously as 2 hour infusion on Day 1 of each cycle. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 16.9 mg: PF-04605412 16.9 mg was administered intravenously as 2 hour infusion on Day 1 of each cycle. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 34 mg: PF-04605412 34 mg was administered intravenously as 2 hour infusion on Day 1 of each cycle. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 68 mg: PF-04605412 68 mg was administered intravenously as 2 hour infusion on Day 1 of each cycle. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 136 mg: PF-04605412 136 mg was administered intravenously as 2 hour infusion on Day 1 of each cycle. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
Period: Overall Study
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Started | 8 | 5 | 3 | 5 | 3 | 9
Completed | 3 | 2 | 2 | 2 | 1 | 1
Not Completed | 5 | 3 | 1 | 3 | 2 | 8
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 4
Not completed — Adverse Event | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease/clinical progression | 0 | 0 | 0 | 3 | 1 | 2
Not completed — Infusion related AEs | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Admission to hospice | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analyzed population is the total number of enrolled subjects who started treatment.
Groups:
- PF-04605412 7.5 mg: PF-04605412 7.5 mg was administered intravenously as 2 hour infusion. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 11.25 mg: PF-04605412 11.25 mg was administered intravenously as 2 hour infusion. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 16.9 mg: PF-04605412 16.9 mg was administered intravenously as 2 hour infusion. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 34 mg: PF-04605412 34 mg was administered intravenously as 2 hour infusion. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 68 mg: PF-04605412 68 mg was administered intravenously as 2 hour infusion. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- PF-04605412 136 mg: PF-04605412 136 mg was administered intravenously as 2 hour infusion. The first cycle lasted 4 weeks and the following cycles lasted 2 weeks each. Treatment was continued until intolerable toxicity, disease progression or participant withdrawal.
- Total: Total of all reporting groups
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg | Total
Number analyzed (Participants) | 8 | 5 | 3 | 5 | 3 | 9 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (10.3) | 54.2 (12.2) | 61.3 (5.5) | 51.8 (7.2) | 60.7 (12.5) | 59.3 (13.6) | 56.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 3 | 1 | 5 | 15
  Male | 4 | 4 | 2 | 2 | 2 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: DLT was defined as any of the following events occurring during the first 28 days of study medication and considered at least possibly-related to study medication: any grade 3 or 4 clinically-relevant non-hematologic toxicity,any >= Grade 3 adverse event (AE) graded by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version 3.0 without a clear alternative explanation to study treatment relationship occurring during the first 6 weeks of treatment with PF-04605412. DLT was used to determine maximum tolerated dose (MTD) in this study.
Time Frame: Baseline up to 6 weeks PF-04605412
Population: All subjects enrolled in the dose escalation part of the study who received at least one dose of study medication that remained on study and/or provided safety follow-up for at least 6 weeks, unless discontinuing due to a DLT. Subjects discontinuing the study due to DLT are included
Measure: Number; unit: participants
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3 | 5
participants | 1 | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: Predose, 1, 2, 2.5, 3, 6, 10, 24 hours after the start of infusion on Day 1; Days 3, 5, 8, 11, 15, 22 of Cycle 1
Population: The analyzed population is all enrolled subjects treated who had received at least 1 dose of PF-04605412 and completed sampling for PK profiles for PF-04605412; N = number of subjects who had reportable Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 7 | 4 | 3 | 4 | 3 | 6
nanogram/milliliter (ng/mL) | 578.3 (37) [lower limit 37] | 1229 (27) [lower limit 27] | 1826 (90) [lower limit 90] | 6682 (11) [lower limit 11] | 13400 (18) [lower limit 18] | 34110 (37) [lower limit 37]

3. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the serum concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: Predose, 1, 2, 2.5, 3, 6, 10, 24 hours after the start of infusion on Day 1; Days 3, 5, 8, 11, 15, 22 of Cycle 1
Population: The analyzed population is all enrolled subjects treated who had received at least 1 dose of PF-04605412 and completed sampling for PK profiles for PF-04605412; N = number of subjects who had reportable AUClast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 7 | 4 | 3 | 4 | 3 | 6
nanogram*hour/milliliter (ng*hr/mL) | 4784 (171) [lower limit 171] | 14440 (170) [lower limit 170] | 12930 (103) [lower limit 103] | 149400 (71) [lower limit 71] | 490600 (85) [lower limit 85] | 2047000 (28) [lower limit 28]

4. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - Inf)]
Description: AUC (0 - inf)= Area under the serum concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Time Frame: Predose, 1, 2, 2.5, 3, 6, 10, 24 hours after the start of infusion on Day 1; Days 3, 5, 8, 11, 15, 22 of Cycle 1
Population: The analyzed population is all enrolled subjects treated who had received at least 1 dose of PF-04605412 and completed sampling for PK profiles for PF-04605412; N = number of subjects who had reportable AUC (0 - inf).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 2 | 0 | 2 | 4 | 3 | 5
ng*hr/mL | 2000 (NA) [lower limit NA] — Geometric mean was not reported for n=<2, instead median was reported |  | 27650 (NA) [lower limit NA] — Geometric mean was not reported for n=<2, instead median was reported | 160600 (69) [lower limit 69] | 505200 (86) [lower limit 86] | 2053000 (28) [lower limit 28]

5. Secondary Outcome: Serum Decay Half-Life (t1/2)
Description: Serum decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Predose, 1, 2, 2.5, 3, 6, 10, 24 hours after the start of infusion on Day 1; Days 3, 5, 8, 11, 15, 22 of Cycle 1
Population: The analyzed population is all enrolled subjects treated who had received at least 1 dose of PF-04605412 and completed sampling for PK profiles for PF-04605412; N = number of subjects who had reportable t1/2.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 2 | 0 | 2 | 4 | 3 | 5
hours | 2.70 (NA) — Mean was not reported for n=<2, instead median was reported |  | 7.27 (NA) — Mean was not reported for n=<2, instead median was reported | 13.5 (3.99) | 19.2 (8.60) | 36.9 (3.96)

6. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax)
Time Frame: Predose, 1, 2, 2.5, 3, 6, 10, 24 hours after the start of infusion on Day 1; Days 3, 5, 8, 11, 15, 22 of Cycle 1
Population: The analyzed population is all enrolled subjects treated who had received at least 1 dose of PF-04605412 and completed sampling for PK profiles for PF-04605412; N = number of subjects who had reportable Tmax.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 7 | 4 | 3 | 4 | 3 | 6
hours | 2.00 [1.00 to 44.7] | 3.04 [3.00 to 5.50] | 2.43 [2.05 to 3.02] | 2.52 [2.00 to 47.4] | 2.00 [2.00 to 2.53] | 6.03 [2.25 to 50.6]

7. Secondary Outcome: Systemic Clearance (CL)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Predose, 1, 2, 2.5, 3, 6, 10, 24 hours after the start of infusion on Day 1; Days 3, 5, 8, 11, 15, 22 of Cycle 1
Population: The analyzed population is all enrolled subjects treated who had received at least 1 dose of PF-04605412 and completed sampling for PK profiles for PF-04605412; N = number of subjects who had reportable CL.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/hr)
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 2 | 0 | 2 | 4 | 3 | 5
Liter/hour (L/hr) | 3.79 (NA) [lower limit NA] — Geometric mean was not reported for n=<2, instead median was reported |  | 0.95 (NA) [lower limit NA] — Geometric mean was not reported for n=<2, instead median was reported | 0.212 (61) [lower limit 61] | 0.135 (58) [lower limit 58] | 0.066 (21) [lower limit 21]

8. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: Predose, 1, 2, 2.5, 3, 6, 10, 24 hours after the start of infusion on Day 1; Days 3, 5, 8, 11, 15, 22 of Cycle 1
Population: The analyzed population is all enrolled subjects treated who had received at least 1 dose of PF-04605412 and completed sampling for PK profiles for PF-04605412; N = number of subjects who had reportable Vss.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 2 | 0 | 2 | 4 | 3 | 5
Liter | 13.65 (NA) [lower limit NA] — Geometric mean was not reported for n=<2, instead median was reported |  | 10.87 (NA) [lower limit NA] — Geometric mean was not reported for n=<2, instead median was reported | 6.61 (66) [lower limit 66] | 5.91 (22) [lower limit 22] | 3.73 (22) [lower limit 22]

9. Secondary Outcome: Number of Participants Positive for Anti-PF04605412 Antibodies
Description: Serum samples were analyzed for anti-drug antibodies (ADA) or human anti-human antibodies (HAHA). This was used to evaluate immunogenicity.
Time Frame: Baseline up to end of treatment
Population: All subjects enrolled in this study who were treated with at least one dose of PF-04605412.
Measure: Number; unit: participants
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 8 | 5 | 3 | 5 | 3 | 9
participants | 1 | 0 | 0 | 0 | 0 | 2

10. Secondary Outcome: Objective Response - Number of Participants With Objective Response
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed responses are those that persist on repeat imaging study ≥4 weeks after initial documentation of response.
  Per RECIST v1.0: CR defined as disappearance of all target lesions and non-target lesions. PR defined as ≥30% decrease in sum of the longest diameters dimensions (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST associated to non-progressive disease response for non target lesions.
Time Frame: Baseline up to 6 weeks after the first infusion of PF-04605412 (end of Cycle 2) and approximately every 6 weeks thereafter only in the absence of progressive disease
Population: All subjects enrolled in this study who were treated with at least one dose of PF-04605412.
Measure: Number; unit: participants
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 8 | 5 | 3 | 5 | 3 | 9
participants | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percent Change in Transfer Constant (Ktrans) From Baseline to Cycle 1 Day 15
Description: Percent change in Ktrans for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) from baseline to Cycle 1 day 15 aimed at defining the effect of PF-04605412 on tumor vasculature.
Time Frame: Screening, and Cycle 1 Day 15
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Percent Change in Initial Area Under the Curve (IAUC)
Description: Percent change in the IAUC for dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) from baseline to Cycle 1 Day 15. IAUC reflects the contrast distribution volume (extravascular extracellular space) in addition to contrast delivery and transport across the vascular endothelium. An IAUC value of zero indicates the absence of disease (ie, no leakage of the contrast agent into the synovial volume); therefore, an increase in this parameter indicates worsening disease (ie, greater permeability of the synovial membrane).
Time Frame: Screening, and Cycle 1 Day 15
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Tissue Macrophage Infiltration
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against tissue macrophages.
Time Frame: Predose and postdose
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Integrin Alpha 5 Beta 1 Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against integrin alpha 5 beta 1.
Time Frame: Predose and postdose
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With CD68 Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies CD68.
Time Frame: Predose and postdose
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Granzyme B Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against Granzyme B.
Time Frame: Predose and postdose
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With CD56 Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against CD56.
Time Frame: Predose and postdose
Population: The analyzed population is all enrolled subjects treated who had received at least 1 dose of PF-04605412 and completed sampling for PK profiles for PF-04605412; N = number of subjects who had reportable CD56 expression.
Measure: Number; unit: Participants
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 7 | 4 | 3 | 5 | 3 | 7
Participants | 6 | 2 | 2 | 3 | 1 | 6

18. Secondary Outcome: Number of Participants With CD16 Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against CD16.
Time Frame: Predose and postdose
Population: The analyzed population is all enrolled subjects treated who had received at least 1 dose of PF-04605412 and completed sampling for PK profiles for PF-04605412; N = number of subjects who had reportable CD16 expression.
Measure: Number; unit: Participants
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 7 | 4 | 3 | 5 | 3 | 7
Participants | 6 | 2 | 2 | 3 | 1 | 6

19. Secondary Outcome: Number of Participants With pFAK Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against pFAK.
Time Frame: Predose and postdose
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With CD31 Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against CD31.
Time Frame: Predose and postdose
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Caspase 3 Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against Caspase 3.
Time Frame: Predose and postdose
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Ki67 Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against Ki67.
Time Frame: Predose and postdose
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Perforin Expression
Description: Immunohistochemical staining of tissue biopsies was performed with monoclonal antibodies directed against Perforin.
Time Frame: Predose and postdose
Population: The data was not statistically analyzed as planned due to early study termination.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04605412 7.5 mg | PF-04605412 11.25 mg | PF-04605412 16.9 mg | PF-04605412 34 mg | PF-04605412 68 mg | PF-04605412 136 mg
Serious Adverse Events (participants affected / at risk) | 5/8 | 2/5 | 1/3 | 1/5 | 0/3 | 5/9
Other Adverse Events (participants affected / at risk) | 8/8 | 5/5 | 3/3 | 4/5 | 3/3 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04605412 7.5 mg (N=8) | PF-04605412 11.25 mg (N=5) | PF-04605412 16.9 mg (N=3) | PF-04605412 34 mg (N=5) | PF-04605412 68 mg (N=3) | PF-04605412 136 mg (N=9)
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Vaginal cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04605412 7.5 mg (N=8) | PF-04605412 11.25 mg (N=5) | PF-04605412 16.9 mg (N=3) | PF-04605412 34 mg (N=5) | PF-04605412 68 mg (N=3) | PF-04605412 136 mg (N=9)
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 1 | 1 | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 5 | 1 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 1 | 2 | 2 | 2 | 3
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 1 | 1 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Prothrombin time (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spider naevus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated prematurely because PK data did not enable sufficient confidence in producing desired clinical benefit. Potential re-occurrence of cytokine mediated infusion reaction at higher doses did not support further development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.